CLINICAL TRIAL: NCT02999945
Title: Body Composition, Metabolic Programming and Long Term Outcome of Growth Restricted Preterm Infants Under Different Nutritional Management A Prospective Randomized Controlled Multicenter Trial
Brief Title: Optimal Growth of Preterm Infants With Growth Restriction
Acronym: OPTIGROW
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding
Sponsor: Medical University of Vienna (Other)
Collaborators: Medical University of Graz (Other); Ludwig-Maximilians - University of Munich (Other); University Hospital Tuebingen (Other); University of Erlangen-Nürnberg Medical School (Other); University of Milan (Other); Poznan University of Medical Sciences (Other); Lund University (Other)
Responsible Party: Principal Investigator, Nadja Haiden,MD, Assoc. Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPTIGROW
Record Dates: First submitted 2016-12-05; First posted 2016-12-21 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Growth Failure; Adiposity; Diabetes; Neurologic Deficits
Keywords: preterm infants; SGA infants; IUGR infants; growth; body composition; metabolomics; microbiome; adiposity markers; metabolic programming; neurodevelopmental outcome
MeSH Terms: conditions — Failure to Thrive; Obesity; Diabetes Mellitus; Neurologic Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SGA-enhanced nutrients (Active Comparator): Infants will receive fortified breast milk (>50% meals/d fortified, 1,4 g protein, 85 kcal/100ml, FM85, Nestle ®) or post discharge formula (2g protein; 73-75 kcal/100ml; Aptamil PDF, Milupa® or Beba F Nestle® ) between discharge and 52nd week of gestation (three months after term)
  Interventions: Dietary Supplement: SGA-enhanced nutrients
- SGA-standard nutrients (Other): Infants will receive unfortified breast milk (65-70kcal/100ml) or starter formula (1,2- 1,3g protein, 66 kcal/100ml Beba Pre Pro Start, Nestle® or Aptamil Pre, Milupa ®) between discharge and 52nd week of gestation (three months after term).
  Interventions: Other: SGA-standard nutrients
- IUGR-enhanced nutrients (Active Comparator): Infants will receive fortified breast milk (>50% meals/d fortified, 1,4 g protein, 85 kcal/100ml, FM85, Nestle ®) or post discharge formula (2g protein; 73-75 kcal/100ml; Aptamil PDF, Milupa® or Beba F Nestle® ) between discharge and 52nd week of gestation (three months after term
  Interventions: Dietary Supplement: IUGR-enhanced nutrients
- IUGR-standard nutrients (Other): Infants will receive unfortified breast milk (65-70kcal/100ml) or starter formula (1,2- 1,3g protein, 66 kcal/100ml Beba Pre Pro Start, Nestle® or Aptamil Pre, Milupa ®) between discharge and 52nd week of gestation (three months after term).
  Interventions: Other: IUGR-standard nutrients

INTERVENTIONS:
Dietary Supplement: SGA-enhanced nutrients — Infants will receive fortified breast milk (>50% meals/d fortified, 1,4 g protein, 85 kcal/100ml, FM85, Nestle ®) or post discharge formula (2g protein; 73-75 kcal/100ml; Aptamil PDF, Milupa® or Beba F Nestle® ) between discharge and 52nd week of gestation (three months after term
  Arms: SGA-enhanced nutrients
Dietary Supplement: IUGR-enhanced nutrients — Infants will receive fortified breast milk (>50% meals/d fortified, 1,4 g protein, 85 kcal/100ml, FM85, Nestle ®) or post discharge formula (2g protein; 73-75 kcal/100ml; Aptamil PDF, Milupa® or Beba F Nestle® ) between discharge and 52nd week of gestation (three months after term
  Arms: IUGR-enhanced nutrients
Other: SGA-standard nutrients — Infants will receive unfortified breast milk (65-70kcal/100ml) or starter formula (1,2- 1,3g protein, 66 kcal/100ml Beba Pre Pro Start, Nestle® or Aptamil Pre, Milupa ®) between discharge and 52nd week of gestation (three months after term)
  Arms: SGA-standard nutrients
Other: IUGR-standard nutrients — Infants will receive unfortified breast milk (65-70kcal/100ml) or starter formula (1,2- 1,3g protein, 66 kcal/100ml Beba Pre Pro Start, Nestle® or Aptamil Pre, Milupa ®) between discharge and 52nd week of gestation (three months after term)
  Arms: IUGR-standard nutrients

SUMMARY:
In this prospective randomized controlled multi center trial the investigators stratify "Very Low Birthweight " (VLBW)-infants with growth retardation in small for gestational age (SGA) or intrauterine growth restricted (IUGR) - infants and aim to investigate the impact of a nutritional management with enhanced nutrients from discharge up to the 52nd week of postconceptional age on growth, body composition, metabolic programming, metabolomics, microbiome and long term neurodevelopmental outcome. In this study, the investigators will evaluate the difference in metabolic profiles of SGA and IUGR preterm infants. The investigators will further longitudinally assess, how different nutritional interventions affect the altered pathways in the first year of life and identify, in combination with data available from metabolic markers, microbiome and breast milk analysis, potential pathways resulting in increased disease risk later in life.

DETAILED DESCRIPTION:
Prematurity is the leading cause for mortality and morbidity in newborns with very low birth weight (VLBW) infants (< 1500g birth weight) at highest risk. Ten to thirty percent of VLBW infants are also born too small for their gestational age defined by a birth weight below the 10th percentile. In daily neonatal intensive care, consequential long term-follow up and most studies all growth restricted premature infants are treated the same, importantly this includes the nutritional management after birth. However, different groups of patients with different causal pathologies are subsumed under the definition growth restriction or born too small. One group of growth restricted patients refers to the infants born constitutionally small or small for gestational age (SGA). The other group refers to infants with an intrauterine growth restriction (IUGR) caused by a complex antenatal pathology. Consequently, the nutritional management after birth is very important to minimize the potential risk for developing obesity, diabetes and cardiovascular diseases later in life and to achieve optimal growth. So far we do not consider the different underlying pathomechanisms of growth restriction in our nutritional concepts for preterm infants and therefore cause long-term consequences. The European society of pediatric gastroenterology, hematology and nutrition (ESPGHAN) recommends to feed enhanced nutrients up to 52nd week of gestation in all growth restricted preterm infants- regardless if they are SGA or IUGR premature. Actually, reliable data guaranteeing that the recommended "enhanced nutrients strategy" providing extra nutrients up to 52 weeks for SGA and IUGR infants is safe and effective for both groups in terms of long-term growth and metabolic programming are lacking.

A total of 348 preterm infants born and discharged below the 10th percentile at term will be included in the study and stratified according to SGA or IUGR by a combination of antenatal ultrasound parameters and growth parameters (including 10% screening failures and 20% drop out. Furthermore IUGR and SGA growth restricted preterm infants will be stratified according to breastfeeding or formula feeding and randomized in one of the following groups: Standard nutrients group (breastfeeding or starter formula) or Enhanced nutrients group (fortified breast milk or post-discharge formula. Body composition measurements will be performed by air displacement plethysmography - a non-invasive method. Anthropometric measurements will be performed by measuring weight, height and head circumference. Furthermore, parameters of metabolic programming, metabolomics, the stool microbiome and neurodevelopmental outcome will be determined. Additionally, the stool microbiome will be characterized from infant stool samples and compared between the two groups. After an interventional period of three months infants will be followed up until 2 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with a birth weight <1500g and birth weight <10th percentile.
* Weight at term <10th percentile
* Informed consent

Exclusion Criteria:

* Genetic or metabolic diseases with the primary effect on growth
* Necrotizing enterocolitis
* Intraventricular hemorrhage (IVH) >Grade II
* Periventricular leukomalacia (PVL) Stage III
* Genetic or metabolic disorders
* Bronchopulmonary dysplasia

Max Age: 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Fat Free Mass | 3 months
  Fat free mass measured by body plethysmography

SECONDARY OUTCOMES:
anthropometry-length | 24 months
  length in cm
anthropometry-weight | 24 months
  weight in grams
anthropometry-HC | 24 months
  head circumference in cm
anthropometry-z-score | 24 months
  z-scores
parameters of metabolic programming- IGF1 | 12 months
  IGF-1in ng/ml
parameters of metabolic programming-IGF3 | 12 months
  IGF-3 in ng/ml
parameters of metabolic programming-IGF-BP | 12 months
  IGF-BP in ng/ml
parameters of metabolic programming-Leptin | 12 months
  Leptin in ng/ml
parameters of metabolic programming-Adiponectin | 12 months
  Adiponectin in mcg/ml
neurodevelopmental outcome | 24months
  Bayley scales
metabolomics | 12 months
  Metabolomic analysis will determine around 200 metabolites covering polar lipids (SOFIA), acylcarnitines (CARN), non-esterified fatty acids (NEFA) and amino acids (AA). Data will be acquired according to retention time and mass transition on triple quadrupole mass spectrometer, controlled by Analyst.
  All metabolite concentrations are reported in µmol/L
stool microbiome | 24 months
macronutrients in breastmilk-fat | 6 months
  Fat will be analysed by modified Mojonnierether extraction (g/100ml)
macronutrients in breastmilk-Lactose | 6 months
  Lactose will be determined by Lactose analysis method: LC-MS/MS (g/100ml)
macronutrients in breastmilk-protein | 6 months
  Protein will be determined by elemental analysis (g/100ml)

CONTACTS AND LOCATIONS:
Overall Officials: Nadja Haiden, MD, Principal Investigator — MUW

IPD SHARING:
Plan to Share IPD: Undecided